CLINICAL TRIAL: NCT00285818
Title: A Double-blind, Placebo-controlled Study of Mifepristone in Patients With Non-psychotic Major Depressive Disorder Referred for Bilateral Electroconvulsive Therapy (ECT)
Brief Title: Mifepristone Treatment for Patients With Non-psychotic Major Depressive Disorder Receiving Bilateral ECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Hugh Brent Solvason, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2HSE450; Oberndorf Family Fund (Other: Stanford University)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2016-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Mifepristone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mifepristone (Active Comparator): Patients receive mifepristone one day before and for 5 additional days after starting ECT
  Interventions: Drug: Mifepristone
- Placebo Oral Capsule (Placebo Comparator): Patients receive a placebo capsule one day before and for 5 additional days after starting ECT
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Mifepristone — Mifepristone is a glucocorticoid receptor antagonist.
  Other Names: RU-486
  Arms: Mifepristone
Drug: Placebo Oral Capsule — Placebo is a capsule without a pharmacological active ingredient
  Other Names: Sugar pill
  Arms: Placebo Oral Capsule

SUMMARY:
The purpose of this study is to see whether the medication mifepristone is an effective and tolerable treatment for increasing the clinical effectiveness of electroconvulsive therapy (ECT) and protecting cognitive function during ECT. Both Mifepristone and ECT appear to normalize hyperfunctioning of the hypothalmic-pituitary-adrenal (HPA) axis, which has been found among patients with major depression referred for ECT. The combination of these two treatments in major depression may lead to a more rapid clinical response than ECT alone. Additionally, there appears to be a connection between pre-ECT higher cortisol levels due to HPA axis hyperfunctioning and post-ECT cognitive impairment. Administration of mifepristone prior to and during ECT treatment may reduce cortisol levels and reduce the incidence of cognitive impairment observed after ECT.

DETAILED DESCRIPTION:
Patients referred to the Stanford ECT Service who provide informed consent for this study will be screened for eligibility.

Day -4 to 0: Screening (visit 1) will occur three to six days prior to the first ECT treatment. Screening procedures will include: Psychiatric interviews and ratings (including MINI, Hamilton Depression Rating Scale and Clinician's Global Impression) and review/retrieval of results of pre-ECT physical exam, ECG, chest x-ray, laboratory evaluations (including comprehensive metabolic panel, comprehensive blood count, and urine toxicology), and vital signs from the subject's medical record. A urine pregnancy test will be included for females of childbearing potential. Concomitant medications and pre-existing health issues will be recorded. Subjects who are deemed eligible for this study will then undergo a battery of neuropsychiatric assessments and will be admitted to GCRC for collection of blood samples to measure adrenocorticotropin (ACTH) and cortisol levels. These samples will be collected hourly beginning at 1pm and ending at 4pm.

Day 1: Subjects will be randomized 1:1 to receive either mifepristone 600mg or placebo each day at bedtime beginning two days prior to the first ECT treatment. Subjects will be administered study medication on Day 1 through Day 8.

Day 3: Subjects will be interviewed with the Hamilton Depression Rating Scale and Clinician's Global Impression before their first ECT treatment.

Day 11: (visit 2) assessments will include psychiatric ratings (including Hamilton Depression Rating Scale and Clinician's Global Impression) and a battery of neuropsychiatric assessments. Adverse events and concomitant medications will be reviewed and recorded. Subjects will be admitted to the GCRC for collection of blood samples to measure ACTH and cortisol levels. Samples will be collected hourly beginning at 1pm and ending at 4pm.

Day 18: (visit 3) assessments will include psychiatric ratings (including Hamilton Depression Rating Scale and Clinician's Global Impression). Adverse events and concomitant medications will be reviewed and recorded. Clinical laboratory assessments will be completed (including a urine pregnancy test for females, comprehensive metabolic panel, comprehensive blood count, urine toxicology, and ECG.) Final visit: (visit 4) will occur 24-72 hours after the last ECT treatment. Assessments will include psychiatric ratings (including Hamilton Depression Rating Scale and Clinician's Global Impression) and a battery of neuropsychiatric assessments. Adverse events and concomitant medications will be reviewed and recorded. A urine pregnancy test will be completed for females.

In addition to the ECT treatment consent, the following materials will be collected from the participant's medical record for every ECT treatment: ECT treatment orders, ECT procedure note and the results of each pre-ECT Montgomery-Asberg Depression Rating Scale (MADRS). ECT treatments at Stanford's ECT Service run every Monday, Wednesday and Friday.

ELIGIBILITY:
Inclusion Criteria:To be considered for participation in the study, subject must meet all of the following criteria:

1. Meets DSM-IV criteria for Major Depressive Episode without psychotic features.

2. 18-75 years of age and able to provide legal consent. 3. Referred to Stanford ECT service by treating physician for bilateral electroconvulsive therapy with inpatient hospitalization.

4. Completed process for consenting to the clinical use of ECT according to California State law.

5. Females of childbearing potential must be using a double-barrier method of contraception during the study and for 30 days after the study (modified 6-2003) Exclusion Criteria:Subjects will be excluded from participation if they meet any of the following criteria:

1. Treatment with ECT in the 6 months prior to screening.
2. Meets criteria for drug or alcohol abuse or dependence in the 6 months prior to screening.
3. Use of alcohol or illegal drugs within seven days of randomization or during study.
4. Presence of unstable or untreated cardiovascular disease, hypertension, or endocrine disorder as determined by investigator.
5. Use of antipsychotic, antidepressant, or other prescription medications unless dose is stable for at least 7 days prior to randomization.
6. Use of any investigational treatment within 30 days of randomization.
7. Current pregnancy.
8. Current lactation.
9. Previous allergic reaction to mifepristone or drugs of similar chemical structure. (added 6-2003)
10. Use of any oral contraceptives or other drugs that may result in adverse drug-mifepristone interaction effects. A 30-day wash out period for oral contraceptives is required before mifepristone begins.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-01; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Brent Solvason, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients receive a placebo capsule one day before and for 5 additional days after starting ECT
  Mifepristone: Mifepristone is a glucocorticoid receptor antagonist.
Period: Overall Study
Arm/Group | Mifepristone | Placebo
Started | 6 | 5
Completed | 2 | 3
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Patients receive a placebo pill one day before and for 5 additional days after starting ECT
  Mifepristone: Mifepristone is a glucocorticoid receptor antagonist.
- Total: Total of all reporting groups
Arm/Group | Mifepristone | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (5.2) | 48.5 (6.2) | 48.3 (5.3)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale Score
Description: The Hamilton Depression Scale measures the severity of depression. There are 17 items rated 0 to 4. A total score of 0 indicates that the patient does not endorse any symptoms of depression. The maximum score (the most severe depression) is 68. The outcome measure is the difference between Visit 1 and Visit 4 Hamilton Depression Rating Scale scores of the mifepristone and placebo groups.
Time Frame: Screening to Final Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Patients receive a placebo pill one day before and for 5 additional days after starting ECT
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 2 | 3
units on a scale
  Baseline | 28.5 (3.9) | 23.0 (5.7)
  Visit 4; 4 weeks | 20.5 (4.9) | 19.0 (7.5)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Mifepristone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 1/6 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=6) | Placebo (N=5)
headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Headache was of mild severity, related to non-specific muscle tension in the temporal and occipital area.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No